CLINICAL TRIAL: NCT00003642
Title: A Phase II Feasibility Study of Combined Accelerated External Radiation and Chemotherapy With 5FU and CDDP Following Transurethral Resection in Patients With Muscle Invasive Transitional Carcinoma of the Bladder - T2-T3, N0, M0 (UICC 1992)
Brief Title: Radiation Therapy and Chemotherapy Following Surgery in Treating Patients With Stage II or Stage III Bladder Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-22971; EORTC-22971
Record Dates: First submitted 1999-11-01; First posted 2004-04-09 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Bladder Cancer
Keywords: stage II bladder cancer; stage III bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Fluorouracil; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of radiation therapy combined with fluorouracil and cisplatin in treating patients who have stage II or stage III bladder cancer, and who have undergone transurethral resection.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the rate of severe acute toxicity occurring during therapy with accelerated external radiotherapy with concurrent fluorouracil (5-FU) and cisplatin following transurethral resection of the bladder in patients with stage II or III muscle invasive transitional cell carcinoma of the bladder. II. Evaluate the rate of freedom from local recurrence to this combined therapy assessed 3 months after the end of treatment in these patients. III. Assess the feasibility of this new therapeutic approach in this patient population. IV. Determine the overall recurrent free survival, long term side effects, and overall survival in these patients.

OUTLINE: This is an open label, multicenter study. Patients undergo accelerated external radiotherapy twice daily 5 days a week for 5 weeks. Concurrent chemotherapy is administered on the first and fifth week consisting of cisplatin IV over 2 hours daily and fluorouracil by 24 hour continuous infusion daily on days 1-5. Patients are followed at 3 months, then every 3 months for the first 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: There will be 19-43 patients accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed unifocal or multifocal transitional cell carcinoma of the bladder no greater than 5 cm, with evidence of muscle invasion documented by transurethral resection of the bladder (TURB), with no residual visible or palpable tumor mass at the end of TURB Stage II or III (T2-T3, N0, M0) No squamous cell or adenocarcinoma No evidence of pelvic lymph node involvement by CT scan or MRI No evidence of hydronephrosis No evidence of distant metastases No disease in the prostatic urethra

PATIENT CHARACTERISTICS: Age: Under 76 Performance status: WHO 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 11 g/dL Hepatic: Not specified Renal: See Disease Characteristics Creatinine clearance greater than 50 mL/min Cardiovascular: No progressive ischemic cardiopathy Other: No reduced bladder capacity No prior or concurrent malignancy except basal cell carcinoma or carcinoma in situ of the cervix treated by hysterectomy

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior immunotherapy for superficial disease allowed No concurrent growth factors Chemotherapy: No prior systemic chemotherapy Prior intravesical chemotherapy or intravesical BCG allowed Endocrine therapy: Not specified Radiotherapy: No prior pelvic radiotherapy Surgery: No prior surgery for bladder cancer except transurethral resection of the bladder

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 1998-10; Primary Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Bolla, MD, Study Chair — CHU de Grenoble - Hopital de la Tronche
Locations (3):
- France (2):
  - Institut Bergonie, Bordeaux
  - CHR de Grenoble - La Tronche, Grenoble
- Dr. Bernard Verbeeten Instituut, Tilburg, Netherlands

REFERENCES:
- [Result] Poortmans PM, Richaud P, Collette L, Ho Goey S, Pierart M, Van Der Hulst M, Bolla M; EORTC Radiation Oncology Group. Results of the phase II EORTC 22971 trial evaluating combined accelerated external radiation and chemotherapy with 5FU and cisplatin in patients with muscle invasive transitional cell carcinoma of the bladder. Acta Oncol. 2008;47(5):937-40. doi: 10.1080/02841860801888799. PMID 18568488